CLINICAL TRIAL: NCT00594321
Title: Evaluation of Fracture Fixation With Energy and Cement in Tumors of the Spine
Acronym: EFFECTS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor closed the trial before it began
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200715482
Record Dates: First submitted 2007-12-21; First posted 2008-01-15 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Spinal Fractures
Keywords: spinal fractures
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Subjects randomized to the control arm of the study will have a standard vertebroplasty with any FDA-approved bone cement done in accordance with the usual method employed by the treating physician.
  Interventions: Device: standard vertebroplasty
- 1 (Experimental): Subjects randomized to the experimental arm of the study will have a vertebroplasty with the SPACE CpsXL Bone cement (FDA-approved) and SPACE 360 Delivery System (FDA-approved).
  Interventions: Device: SPACE CpsXL Bone Cement and SPACE 360 Delivery System

INTERVENTIONS:
Device: SPACE CpsXL Bone Cement and SPACE 360 Delivery System — SPACE CpsXL Bone Cement and SPACE 360 Delivery System
  Arms: 1
Device: standard vertebroplasty — standard vertebroplasty
  Arms: 2

SUMMARY:
The objective of the clinical trial is to evaluate the SPACE 360 Delivery System using SPACE CpsXL Bone Cement compared to standard vertebroplasty in the treatment of pathological fractures of the spine caused by metastatic tumors of the spine, myeloma, or lymphoma. Up to a total of three levels per patient may be included or five levels for multiple myeloma. The control group will be standard vertebroplasty.

DETAILED DESCRIPTION:
The primary endpoint is cement leakage as determined radiographically (CT). will be cement leakage measured by CT. Secondary endpoints are reduction of pain (VAS) and quality of life measurements (Oswestry disability index).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 85 years of age
2. Pain at one to three levels, or five for multiple myeloma (pain on palpation/percussion over fractured vertebral body) requiring treatment
3. Spinal metastasis (except renal cell), myeloma, or lymphoma of the spine
4. Pathological fracture(s), T5-L5, with bone marrow edema imaged by magnetic resonance imaging (MRI)
5. Visual Analog Scale (VAS) for pain of > 4 on a scale of 0 to 10
6. Oswestry score of at least a moderate disability (21-40%)
7. No major surgery to the spine planned for at least 1 month following enrollment - Defined as a procedure the magnitude of a laminectomy or more
8. Life expectancy of > 6 months.
9. Patient has sufficient mental capacity to comply with the protocol requirements
10. Availability for all study visits and phone calls
11. Understands the potential risks and benefits of participating in the study and is willing to provide written informed consent
12. Pathological vertebral fracture with 20-70% compression (compared to adjacent normal vertebral body)
13. Fracture age < 6 months
14. Signal on MRI consistent with non-healed fracture
15. Female subjects must either be no longer capable of reproduction or taking acceptable measures to prevent pregnancy during the study
16. Subject must be willing and able to comply with specified follow-up evaluations

Exclusion Criteria:

1. Primary tumors other than plasmacytoma
2. Renal cell tumors
3. More than 80% compression of the vertebrae
4. Level(s) above T7 to treat
5. Fractures due osteoporosis
6. Burst fracture
7. Pedicle fracture
8. Neurological deficit associated with the fracture
9. Kyphosis > 30°
10. Translation > 4 mm
11. Instability of posterior wall with symptomatic displacement of fragment into spinal canal or significant canal compromise
12. Intercostal nerve compression
13. Active systemic or local infection at the level(s) to be treated
14. Myelopathy
15. Uncontrolled coagulopathy
16. Cannot temporarily discontinue anticoagulation therapy
17. Known allergy to device materials / PMMA
18. Radiculopathy
19. Cord compression or canal compromise requiring surgery for decompression
20. High energy trauma
21. Severe cardiopulmonary deficiencies - Defined as not being able to tolerate general anesthesia (although the likelihood is local anesthesia will be used)
22. Vertebra plana defined as vertebral body height of 20% or less compared to the nearest normal level
23. Disabling back pain secondary to another cause that may interfere with accurate data collection
24. Subjects who are known to be pregnant (pregnancy test required within 10 days of treatment) or lactating
25. Females capable of reproduction and will not take acceptable measures to prevent reproduction during the study
26. Subjects who test positive for HIV
27. Currently enrolled in another investigational device trial (IDE) that has not completed the protocol required primary follow-up period (excludes 15 year follow-up of gene therapy trials)
28. Lesions involving the pedicle
29. Platelet count of < 50,000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is cement leakage as determined radiographically (CT). will be cement leakage measured by CT. | 3 years

SECONDARY OUTCOMES:
Secondary endpoints are reduction of pain (VAS) and quality of life measurements (Oswestry disability index). | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Arthur B. Dublin, M.D., Principal Investigator — UC Davis Dept. of Radiology
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States